CLINICAL TRIAL: NCT00675350
Title: A Pharmacokinetic Study of Homoharringtonine (Omacetaxine Mepesuccinate) Administered Subcutaneously to Patients With Advanced Solid and Hematologic Tumors
Brief Title: Pharmacokinetic (PK) Study of Homoharringtonine (Omacetaxine Mepesuccinate) Administered Subcutaneously to Patients With Advanced Solid and Hematologic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ChemGenex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CGX-635-205
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Hematologic Tumors
Keywords: Omacetaxine; Homoharringtonine; HHT; Solid and hematologic malignant tumors
MeSH Terms: interventions — Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Homoharringtonine (Experimental)
  Interventions: Drug: Omacetaxine

INTERVENTIONS:
Drug: Omacetaxine — 1.25 mg/m2 subcutaneous twice daily for 14 days
  Other Names: Homoharringtonine; HHT

SUMMARY:
PK Study of Homoharringtonine (Omacetaxine Mepesuccinate) Administered Subcutaneously to Patients With Advanced Solid and Hematologic Tumors

DETAILED DESCRIPTION:
This is an open-label non-randomized pharmacokinetic (PK) study of Homoharringtonine (Omacetaxine Mepesuccinate) administered as a subcutaneous (SC)injection to patients with relapsed and/or refractory hematologic malignancies and to patients with advanced solid tumors with no bone marrow involvement.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years old.
* Be diagnosed with relapsed or refractory leukemia including chronic myelogenous leukemia (CML), acute promyelocytic leukemia (APL), acute myelogenous leukemia (AML), or myelodysplastic syndrome (MDS)

  * Relapsed defined as reappearance of leukemic blasts in the peripheral blood or the finding of ≥5% blasts in the bone marrow, not attributable to another cause (e.g., bone marrow regeneration after consolidation therapy).
  * Refractory defined as no response to previous combined chemotherapy regimens including at least one cytarabine plus one anthracycline advanced solid tumors (i.e., breast, lung, head / neck, colorectal, melanoma, and sarcoma). Patients must have exhausted or become intolerant to all available therapies.
* (Patients with hematologic malignancies): Have completed all previous anti-leukemic therapy (except leukapheresis) at least 2 weeks prior to the first planned dose of OMA and must have fully recovered from side effects of a previous therapy unless, disease progression necessitates early therapy. Leukapheresis is allowed up to 24 hours prior to registration.
* (Patients with solid tumors): Patients may have measurable or unmeasurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional computerized tomography (CT) or magnetic resonance imaging (MRI) scans, or as ≥10 mm with spiral computerized tomography (CT) scan. Imaging must be performed within 28 days of the first dose of study drug.
* Have an estimated life expectancy of ≥12 weeks
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2 (see Appendix B)
* Be able to provide written informed consent prior to enrollment into the study. In the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed.
* Be male or a non-pregnant, non-lactating female. Fertile patients must agree to use an effective barrier method contraception (e.g., latex condom, diaphragm, or cervical cap) to avoid pregnancy while on therapy and for 6 months following the discontinuation of the study drug.
* A non-fertile female is defined as:

  * Postmenopausal (amenorrheic for ≥12 months) Undergone a complete oophorectomy or hysterectomy.
* Have a negative serum pregnancy test within 7 days prior to the first dose of study drug (if patient is a female of childbearing potential).
* QTc <450 ms on screening 12-lead ECG (using Bazett's correction of QT interval formula [QTcB]).
* Have adequate organ function as indicated by the following laboratory values obtained within 7 days prior to the first dose of study drug as outlined in Table 3.
* Be able and willing to comply with the requirements of the entire study.

Exclusion Criteria:

* Received previous treatment with OMA within 6 months of study entry.
* Have New York Heart Association (NYHA) Class 3 or 4 heart disease, active ischemia, or any uncontrolled, unstable cardiac condition for which treatment for the condition is indicated but is not controlled despite adequate therapy, including angina pectoris, cardiac arrhythmia, hypertension, or congestive heart failure (see Appendix D).
* Experienced a myocardial infarction in the previous 12 weeks.
* Have solid tumors with known bone marrow or central nervous system (CNS) involvement.
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Are pregnant or lactating.
* Received systemic chemotherapy in the 4 weeks prior to first dose of study drug, unless treatment is required for progressive leukemia. In patients with rapidly proliferating disease, hydroxyurea may be administered immediately prior to and during the first two cycles of treatment, if clinically indicated, to control disease.
* Received radiation therapy within 6 weeks of the first dose of study drug. Localized radiation for palliation may be administered with 2 weeks of the first dose of study drug.
* Have any medical condition or psychiatric disorder(s) rendering the patient unable to understand the nature, scope, and possible consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Evaluation | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, M.D., Principal Investigator — Mary Crowley Cancer Research Center
Locations (1):
- Mary Crowley Cancer Research Center, Dallas, Texas, United States